CLINICAL TRIAL: NCT01650116
Title: Evaluation of Sodium Urinary Excretion, Chlorine Urinary Excretion, Urinary Partial CO2 Pressure as Renal Perfusion Indicators During Liver Transplant. Comparison With Other Polemic State Indicators (Such as PiCCO, ScvO2, O2 Delivery).
Brief Title: Evaluation of Hemodynamics and Amount of Blood Flowing Through the Kidneys During Liver Transplant by Measuring Some Physiological Substances in Blood and Urines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Dr. Paolo Feltracco, Principal Investigator, Azienda Ospedaliera di Padova
Other Study IDs: 2661P
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Hypovolemia During Liver Transplantation; Renal Hypoperfusion During Liver Transplantation
Keywords: hypovolemia; renal hypoperfusion; liver transplantation; sodium; chloride; PuCO2; ScvO2; PiCCO; O2-delivery; hemodynamic indexes
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to verify any existing relationship between urinary parameters (such as excretion of sodium, chlorine, urinary partial CO2 pressure [PuCO2]) and general volemic indicators (such as PiCCO, ScvO2, O2 delivery) during liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* surgery for liver transplantation
* age 18-75
* ASA class I-III

Exclusion Criteria:

* age above 75 or under 18
* ASA class IV
* pre-existing renal failure
* pregnant patients
* patients unable to give written consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Determination of hemodynamic indicators (PiCCO, ScvO2, O2-delivery) and three urinary analytes (sodium, chloride, CO2 partial pressure) | During the stay of the patient in the operating room (in average 8 hours) and the subsequent stay in the post-surgery intensive care unit (in average 5 days)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Ori, Prof. M.D., Study Chair — Università degli Studi di Padova - Azienda Ospedaliera di Padova; Paolo Feltracco, M.D., Principal Investigator — Azienda Ospedaliera di Padova; Andrea Bortolato, M.D., Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, Padova, Italy